CLINICAL TRIAL: NCT06349057
Title: Anticholinergic Burden as a Modifiable Risk Factor in Cardiac Surgery: Evidence From a Randomized Controlled Study
Brief Title: The Effect of the Anticholinergic Burden Following Elective Coronary Artery Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Muhammed Çobas, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AnkaraCHBilkent.1
Record Dates: First submitted 2024-03-17; First posted 2024-04-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Recovery; Length of Hospital Stay; Postoperative Complications
Keywords: cardiac surgery; anticholinergic burden; elderly; represcribing
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): There will be no intervention in the perioperative period, data will be collected only by observation. Anesthesia management, surgical procedure and postoperative care will be applied as routine.
- Remifentanyl, Propofol, Sevoflurane / Desflurane, Propofol (Active Comparator): Preoperative period : There will be no intervention.
  Intraoperative period : An erector spinae plane block will be applied before anesthesia induction. Drugs with cholinergic burden will not be preferred. Lower anticholinergic drugs will be used. There will be no intervention in the surgical procedure.
  Postoperative period : Drugs with high cholinergic burden will not be used. Lower anticholinergic drugs will be used.
  Intraoperative and postoperative periods, instead of drugs with high anticholinergic burden; lower burden drugs will be preferred.
  High anticholinergic burden drugs: (Fentanyl -, Tramadol-, Midazolam , Pancuronium9
  Lower burden drugs : (Remifentanyl, Sevoflurane, Desflurane, Propofol, Rocuronium, Lidocaine)
  Interventions: Drug: reducing anticholinergic burden

INTERVENTIONS:
Drug: reducing anticholinergic burden — In the intraoperative and postoperative periods instead of drugs with high anticholinergic burden; drugs with low burden will be preferred.
  Other Names: not reducing anticholinergic burden, routine care
  Arms: Remifentanyl, Propofol, Sevoflurane / Desflurane, Propofol

SUMMARY:
Anticholinergic drugs are common in older adults and linked to cognitive decline, frailty, longer hospital stay, and higher mortality. This cumulative burden, often increased by anesthetics and analgesics, may worsen during surgery. The study evaluates whether reducing perioperative anticholinergic load improves recovery after cardiac surgery.

DETAILED DESCRIPTION:
Anticholinergic agents are frequently prescribed in older adults and have been linked to negative outcomes such as cognitive decline, frailty, extended hospitalization, and increased mortality. The cumulative exposure, referred to as anticholinergic burden, may be exacerbated during the perioperative period due to anesthetic and analgesic use. This trial explores whether minimizing perioperative anticholinergic burden can improve postoperative recovery following cardiac surgery. In this prospective, randomized controlled study, 120 patients aged 60 years or older undergoing isolated coronary artery bypass grafting with a preoperative Anticholinergic Cognitive Burden score of ≥3 were included. Participants were assigned either to standard perioperative care involving anesthetic and analgesic agents with anticholinergic activity (Group Standard) or to a deprescribing protocol excluding all anticholinergic drugs intraoperatively and postoperatively (Group Deprescribing). The primary endpoints were functional recovery assessed at 90 days using the Katz Index and Clinical Frailty Scale. Secondary endpoints comprised hospital length of stay, 90-day incidence of cardiac and pulmonary complications, intensive care Unit stay, duration of mechanical ventilation, additional complications, and 90-day mortality. The Wilcoxon signed-rank test was used for paired comparisons of Katz and frailty scores, while multivariate logistic regression was applied to identify independent predictors of postoperative cardiac complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary artery bypass surgery
* Patients with high anticholinergic burden

Exclusion Criteria:

* All other procedures except isolated coronary bypass surgery
* Patients with low anticholinergic burden
* Patients whose records cannot be accessed through the data system

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Katz Index of Independence in Activities of Daily Living and Clinical Frailty Scale (CFS) | Postoperative day 90
  The Katz Index of Independence in Activities of Daily Living evaluates a patient's ability to perform six basic functions: bathing, dressing, toileting, transferring, continence, and feeding. Each activity is scored as either "independent" (1 point) or "dependent" (0 points). The total score reflects the patient's overall level of functional independence.
  The Clinical Frailty Scale (CFS) is a validated 9-point tool used to assess a patient's baseline frailty status. It evaluates physical fitness, comorbidity burden, functional dependence, and overall health status. Scores range from 1 (Very Fit) to 9 (Terminally Ill). Higher scores indicate greater frailty and worse baseline physiological reserve.

SECONDARY OUTCOMES:
Intensive Care Unit Length of Stay (days) | From postoperative ICU admission until ICU discharge (typically within 1-3 days).
  The duration of stay in the intensive care unit, measured in days, from ICU admission after surgery until ICU discharge.
Duration of Mechanical Ventilation (hours) | From the end of surgery to extubation
  The duration of postoperative mechanical ventilation, measured in hours, from end of surgery until successful extubation.
other postoperative complications | From completion of surgery to postoperative day 90
  Occurrence of postoperative complications within 90 days after surgery, including neurological (stroke, transient ischemic attack, seizures), renal (acute kidney injury, need for renal replacement therapy, chronic renal failure), and infectious complications (pneumonia, mediastinitis, meningitis, urinary tract infection, wound infection, catheter-related sepsis), as well as delirium.
all-cause mortality | From completion of surgery to postoperative day 90
  All-cause mortality occurring within 90 days after surgery.
Change in Katz Index of Independence in Activities of Daily Living From Baseline | Baseline (preoperative) to postoperative day 90
  The change in Katz Index score will be calculated as the postoperative day 90 score minus the preoperative baseline score. The Katz Index ranges from 0 (highly dependent) to 6 (independent). Higher scores indicate better functional independence.
Postoperative major cardiac complications | From completion of surgery to postoperative day 90
  Incidence of major postoperative cardiac complications, including cardiac arrest, myocardial infarction, arrhythmia, and aortic dissection.
Hospital length of stay (days) | From hospital admission for surgery until hospital discharge (typically within 5-10 days).
  Duration of postoperative hospital stay, measured in days, from admission to the hospital after surgery until hospital discharge.
Incidence of major pulmonary complications | From completion of surgery to postoperative day 90
  Major postoperative pulmonary complications, including pneumothorax, pleural effusion, pulmonary embolism, and acute respiratory distress syndrome (ARDS).
Change in Clinical Frailty Scale (CFS) from baseline | Baseline (preoperative) to postoperative day 90
  Change in Clinical Frailty Scale (CFS) score from preoperative baseline to postoperative day 90.
  The CFS is a nine-point scale assessing mobility, energy, physical activity, and overall functional health:
  1. = Very Fit
  2. = Well
  3. = Managing Well
  4. = Vulnerable
  5. = Mildly Frail
  6. = Moderately Frail
  7. = Severely Frail
  8. = Very Severely Frail
  9. = Terminally Ill Higher scores indicate greater frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Aykut, specialist, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Aslihan Aykut, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hebert M, Cartier R, Dagenais F, Langlois Y, Coutu M, Noiseux N, El-Hamamsy I, Stevens LM. Standardizing Postoperative Complications-Validating the Clavien-Dindo Complications Classification in Cardiac Surgery. Semin Thorac Cardiovasc Surg. 2021 Summer;33(2):443-451. doi: 10.1053/j.semtcvs.2020.09.029. Epub 2020 Sep 24. PMID 32979483
- [Result] Salahudeen MS, Hilmer SN, Nishtala PS. Comparison of anticholinergic risk scales and associations with adverse health outcomes in older people. J Am Geriatr Soc. 2015 Jan;63(1):85-90. doi: 10.1111/jgs.13206. PMID 25597560
- [Result] Magin PJ, Morgan S, Tapley A, McCowan C, Parkinson L, Henderson KM, Muth C, Hammer MS, Pond D, Mate KE, Spike NA, McArthur LA, van Driel ML. Anticholinergic medicines in an older primary care population: a cross-sectional analysis of medicines' levels of anticholinergic activity and clinical indications. J Clin Pharm Ther. 2016 Oct;41(5):486-92. doi: 10.1111/jcpt.12413. Epub 2016 Jun 27. PMID 27349795